CLINICAL TRIAL: NCT00501943
Title: Neuroprotection With Riluzole in Patients With Early Multiple Sclerosis
Brief Title: Neuroprotection With Riluzole Patients With Early Multiple Sclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Multiple Sclerosis Society (Other); Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Emmanuelle Waubant, Associate Professor of Clinical Neurology, University of California, San Francisco
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: H9924-29155-05
Record Dates: First submitted 2007-07-12; First posted 2007-07-16 (Estimated); Results first posted 2014-04-09 (Estimated); Last update posted 2014-04-09 (Estimated); Status verified 2014-03

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Interferon beta-1a; Riluzole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Riluzole (Active Comparator): Riluzole + Avonex
  Interventions: Drug: Avonex (Interferon beta 1a); Drug: Riluzole
- Placebo (Placebo Comparator): placebo + Avonex
  Interventions: Drug: Avonex (Interferon beta 1a); Drug: Placebo

INTERVENTIONS:
Drug: Avonex (Interferon beta 1a)
Drug: Riluzole
  Arms: Riluzole
Drug: Placebo
  Arms: Placebo

SUMMARY:
This is a double blind, randomized, parallel group design placebo-controlled mono-center study. Patients will be evaluated within twelve months of CIS onset. Patients with at least 2 silent ovoid T2 bright areas in the deep white matter on their clinic brain MRI scan will be offered participation in the study. Patients will be randomized to oral riluzole or placebo (1:1). Patient will take 50 mg of riluzole or placebo once a day for one month. If 50 mg once a day is well tolerated, patients will then go on 50 mg twice daily for the rest of the study. They will start Avonex (Interferon beta 1a) therapy 30 mcg IM once weekly 3 months after study drug (riluzole or placebo) is initiated if their liver function has remained normal.

Forty patients within twelve months of onset CIS onset will be enrolled at UCSF MS Center. Patients will be evaluated every month for the first 12 months and every three months thereafter for a total study duration of 24-month. Enrollment period will last six months.

DETAILED DESCRIPTION:
To determine the effect of riluzole up to 50 mg bid on MRI parameters, including T1 lesions load, atrophy of gray and white matter, and 1H-MRSI; and to determine safety of riluzole when administered orally up to 50 mg bid for 2 years in double blinded clinical trial of patients with clinically isolated syndromes (CIS) and at least 2 silent T2-bright areas in the deep white matter. These patients have a high risk of conversion to MS within 2 years and faster rate of atrophy (Dalton 2004).

Specific aims:

1. To determine the effect of treatment compared to placebo on annual change in measures of normalized brain gray and white matter volume changes.
2. To determine the effect of riluzole compared to placebo on annual change in proton spectroscopic intensities of N-acetyl aspartate (NAA) and glutamate in normal appearing white matter (NAWM), in acute and chronic lesions.
3. To determine the safety of riluzole up to 50 mg bid in patients with CIS in association to Avonex (Interferon beta 1a) 30 mcg IM once a week.
4. To monitor changes on MS functional composite (MSFC) (Cutter 1999, Rudick 1998), optic coherence tomography (OCT), low contrast sensitivity and EDSS in these patients.
5. To monitor recovery from exacerbations.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must give written informed consent;
2. Patients with a early MS or clinically isolated syndromes (CIS) in the past 12 months as defined by an acute or sub-acute episode suggestive of demyelination affecting the optic nerves, brain stem or spinal cord or other central nervous system location.
3. Entry age 18-55
4. Males and females
5. At least 2 silent T2 bright areas in the deep white matter on screening brain MRI.
6. No riluzole, interferon, copaxone, cyclophosphamide, mitoxantrone or other off-label immunosuppressive drugs for MS prior to study entry
7. No corticosteroid during the 4 weeks prior to baseline MRI exam
8. No prior exposure to total lymphoid irradiation
9. No history of substance abuse, including documented alcohol dependence within 6 months prior to screening or alcohol liver damage with AST , ALT > twice upper normal limits
10. No pregnant or nursing patients
11. No history of systemic illness or medical condition that would limit the likelihood of completing the gadolinium-enhanced MRI procedures. Automatic exclusionary conditions will include hypersensitivity reaction to riluzole or any of the tablets components, uncontrolled hypertension, epilepsy, and insulin dependent diabetes, asthma, known malignancy other than skin cancer, symptomatic cardiac disease or metallic objects on or inside the body.
12. Patients willing to use birth control during the study.
13. Patients willing to go on Avonex therapy 3 months after being randomized to study drug and no contra-indication to use of interferon therapy.

Exclusion Criteria:

1. A history of major depression or psychosis.
2. A clinically significant MS exacerbation within 30 days of the screening
3. Pregnancy
4. Abnormal screening liver function (AST or ALT > twice the upper normal limit).
5. Patients receiving hepatotoxic medications such as drugs interfering with CYP 1A2.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2006-07; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuelle Waubant, MD, PhD, Principal Investigator — UCSF , MS Center; Emmanuelle Waubant, MD PhD, Principal Investigator — UCSF, MS Center
Locations (1):
- UCSF MS Center , 675 Nelson Rising Lane, Suite 221, San Francisco, California, United States

REFERENCES:
- [Derived] Kuhle J, Nourbakhsh B, Grant D, Morant S, Barro C, Yaldizli O, Pelletier D, Giovannoni G, Waubant E, Gnanapavan S. Serum neurofilament is associated with progression of brain atrophy and disability in early MS. Neurology. 2017 Feb 28;88(9):826-831. doi: 10.1212/WNL.0000000000003653. Epub 2017 Feb 1. PMID 28148632
- [Derived] Maghzi AH, Graves J, Revirajan N, Spain R, Liu S, McCulloch CE, Pelletier D, Green AJ, Waubant E. Retinal axonal loss in very early stages of multiple sclerosis. Eur J Neurol. 2015 Jul;22(7):1138-41. doi: 10.1111/ene.12722. Epub 2015 Apr 29. PMID 25929276

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with diagnosis of early Relapsing Remitting MS were invited to participate in the study at 2 US sites- UCSF and OHSU during the period between Dec 2007 and May 2010
Groups:
- Riluzole: Riluzole
  Riluzole 50 mg BID added to weekly injection of Interferon beta 1a
- Placebo: placebo
  1 tab of Placebo BID added to weekly injection of Interferon beta 1a
Period: Overall Study
Arm/Group | Riluzole | Placebo
Started | 22 | 21
Completed | 20 | 18
Not Completed | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Riluzole | Placebo | Total
Number analyzed (Participants) | 22 | 21 | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.2 (9.84) | 32.4 (7.85) | 36 (9.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 14 | 31
  Male | 5 | 7 | 12
Region of Enrollment [Number; unit: participants]
  United States | 22 | 21 | 43

OUTCOME MEASURES:

1. Primary Outcome: MRI Parameter- Percent Brain Volume Change for 2 Years
Description: Baseline MRI is compared to MRI images collected during subsequent timepoints. The percent brain volume change is measured using SIENAX (Structural Image Evaluation using Normalization of Atrophy-X)
Time Frame: Baseline, Month-3, Month-6, Month-12, Month-18 and Month-24
Population: Multivariate regression model was used as the statistical method of analysis for the study. So data from patients who have not completed the study are also used for statistical analysis.
Measure: Mean (95% Confidence Interval); unit: percent change per year
Arm/Group | Riluzole | Placebo
Number analyzed (Participants) | 22 | 21
percent change per year | -0.862 [-1.168 to -0.556] | -0.49 [-0.766 to -0.208]

2. Secondary Outcome: Changes in Normalized White Matter Volumes (nWMV)
Description: The baseline data of white matter volume obtained from the MRI images is compared to data obtained at time points using SIENA (Structural Image Evaluation using Normalization of Atrophy) and SIENAX
Time Frame: Baseline, Month-3, Month-6, Month-12, Month-18 and Month-24
Measure: Mean (95% Confidence Interval); unit: percent change per year
Groups:
- Riluzole: Riluzole
  Riluzole or Placebo, and Avonex(Interferon beta 1a): Riluzole, Placebo and Avonex(Interferon beta 1a)
- Placebo: placebo
  Riluzole or Placebo, and Avonex(Interferon beta 1a): Riluzole, Placebo and Avonex(Interferon beta 1a)
Arm/Group | Riluzole | Placebo
Number analyzed (Participants) | 22 | 21
percent change per year | -1.75 [-14.709 to 11.213] | -9.69 [-22.206 to 2.825]

3. Secondary Outcome: Changes in MS Functional Composite (MSFC)
Description: Baseline MSFC data is compared to MSFC data collected during the timepoints. The MSFC is a three-part, standardized, quantitative, assessment instrument that measures the clinical dimensions of leg function, arm/hand function and cognitive function and the components include Timed 25-Foot walk, 9-Hole Peg Test and Paced Auditory Serial Addition Test.
Time Frame: Baseline, Month-3, Month-6, Month-12, Month-18 and Month-24
Measure: Mean (95% Confidence Interval); unit: percent change per year
Arm/Group | Riluzole | Placebo
Number analyzed (Participants) | 22 | 21
percent change per year | 0.041 [-0.043 to 0.126] | 0.052 [-0.030 to 0.133]

4. Secondary Outcome: Changes in Peripapillary Retinal Nerve Fiber Layer Thickness (RNFL)
Description: Baseline RNFL data is compared to the RNFL data collected during the timepoint, and the changes in RNFL is measured using optical coherence tomography (OCT).
Time Frame: Baseline, Month-3, Month-6, Month-12, Month-18 and Month-24
Measure: Mean (95% Confidence Interval); unit: percent change per year
Arm/Group | Riluzole | Placebo
Number analyzed (Participants) | 22 | 21
percent change per year | -4.670 [-9.309 to -0.032] | -1.839 [-6.692 to 3.014]

5. Secondary Outcome: Changes in Symbol Digit Modality Test (SDMT)
Description: Baseline SDMT data were compared to SDMT data collected during the timepoints. A simple substitution task, the SDMT gives the examinee 90 seconds to pair specific numbers with given geometric figures as a measure for screening cognitive impairment. The total score is the total number of correctly completed boxes in the time allowed. The test score range is from 0(worst outcome) to 110 (best outcome).
Time Frame: Baseline, Month-3, Month-6, Month-12, Month-18 and Month-24
Measure: Mean (95% Confidence Interval); unit: percent change per year
Arm/Group | Riluzole | Placebo
Number analyzed (Participants) | 22 | 21
percent change per year | 0.342 [-0.774 to 1.457] | 0.417 [-0.703 to 1.537]

6. Secondary Outcome: Changes in Normalized Grey Matter Volume
Description: The baseline data of grey matter volume obtained from the MRI images is compared to data obtained at time points using SIENA (Structural Image Evaluation using Normalization of Atrophy) and SIENAX
Time Frame: Baseline, Month-3, Month-6, Month-12 and Month-24
Measure: Mean (95% Confidence Interval); unit: percent change per year
Arm/Group | Riluzole | Placebo
Number analyzed (Participants) | 22 | 21
percent change per year | -14.369 [-30.566 to 1.827] | -18.444 [-34.434 to -2.454]

ADVERSE EVENTS:
Time Frame: From screening to Month-24 / withdrawal visit.
Arm/Group | Riluzole | Placebo
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/21
Other Adverse Events (participants affected / at risk) | 15/22 | 15/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Riluzole (N=22) | Placebo (N=21)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 7 (7)
dizziness (Ear and labyrinth disorders) | 9 (9) | 5 (5)
Elevated liver function tests (Hepatobiliary disorders) | 2 (2) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes